CLINICAL TRIAL: NCT02268136
Title: A Single-blind, Placebo-controlled, Parallel Group, Single Increasing Dose Tolerance Study in Healthy Male Volunteers After Intravenous Administration of BIII 890 CL (Dosage: 0.5 mg/h - 80 mg/h), Infusion Time 1 Hour.
Brief Title: Increasing Dose Tolerance Study in Healthy Male Volunteers After Administration of BIII 890 CL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 599.1
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — BIII 890 CL

ARMS (2):
- BIII 890 CL (Experimental): single increasing doses
  Interventions: Drug: BIII 890 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIII 890 CL
  Arms: BIII 890 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective ot the present study is to obtain information about safety, tolerability and preliminary pharmacokinetics of BIII 890 CL after single intravenous administration of increasing doses in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Age ≥ 21 and ≤ 50 years
* Broca index ≥ - 20% and ≤ + 20%
* Signed written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Results of the medical examination, laboratory tests or electrocardiogram recordings are judged by the clinical investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy), central nervous system trauma in the medical history or with psychiatric disorders or neurological disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (≥ 24 hours) within the last month or less than ten half-lives of the respective drug before enrolment in the study
* Intake of any other drugs which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smokers (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Volunteers who are not able to refrain from smoking on study days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Participation in excessive physical activities (e.g. competitive sports) within the last week before the study
* Blood donation (≥ 100 ml) within the last 4 weeks

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 1999-04; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically relevant changes in vital signs | up to 8 days after drug administration
Number of subjects with adverse events | up to 8 days after drug administration
Number of subjects with clinically relevant changes in electrocardiogram | up to 8 days after drug administration
Number of subjects with clinically relevant changes in pharmaco electroencephalogram (EEG) | up to 24 hours after drug administration
Number of subjects with clinically relevant changes in laboratory parameters | up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 24 hours after drug administration
Time to reach Cmax (tmax) | up to 24 hours after drug administration
Terminal half-life (t1/2) | up to 24 hours after drug administration
Area under the plasma concentration-time curve (AUC) for several time points | up to 24 hours after drug administration
Mean residence time (MRT) | up to 24 hours after drug administration
Plasma clearance (CL) | up to 24 hours after drug administration
Volume of distribution (Vz) | up to 24 hours after drug administration
Amount of the analyte excreted in urine (Ae) | up to 24 hours after drug administration